CLINICAL TRIAL: NCT01463410
Title: Accuracy Testing of the Chromosomal Aberration and Gene Mutation Markers of the AMLProfiler
Status: Terminated | Type: Observational
Why Stopped: The required number of banked samples could not be met due to limited availability. There is no realistic possibility to complete the study succesfully.
Sponsor: Skyline Diagnostics BV (Industry)
Collaborators: Illumina, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PROT-015
Record Dates: First submitted 2011-10-28; First posted 2011-11-01 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Promyelocytic Leukemia (APL); Refractory Anemia With Excess of Blasts (RAEB)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — RNA from bone marrow samples will be retained.
Oversight: Data Monitoring Committee: No

SUMMARY:
This clinical study will demonstrate the accuracy of the chromosomal aberration and gene mutation markers of the AMLProfiler molecular diagnostic assay and generate clinical performance data to support a Pre-Market Approval (PMA) submission to the Food and Drug Administration for in vitro diagnostic use within the United States of America.

The objective is to demonstrate the positive and negative percent agreement of each marker by comparing AMLProfiler results from multiple clinical participating sites with data generated using a laboratory developed bi-directional sequencing method generated at the molecular diagnostic reference lab.

The AMLProfiler assay is a qualitative in vitro diagnostic test for the detection of AML or APL specific chromosomal aberrations (specific recurrent translocations and inversions), as well as expression of specific genetic markers in RNA extracted from bone marrow aspirates of patients with Acute Myeloid Leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a cytopathologically confirmed diagnosis of AML subjects with refractory anemia with excess of blasts (RAEB) according to the WHO 2008 classification
2. ≥ 18 years
3. Written informed consent

Exclusion Criteria:

1. Subjects without a cytopathologically confirmed diagnosis of AML subjects with refractory anemia with excess of blasts (RAEB) according to the WHO 2008 classification
2. < 18 years
3. Without written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bone marrow samples will be used in the study only from AML,APL or RAEB subjects. Written informed consent by subjects will be obtained for use of their bone marrow samples in this study. Each site will follow their own bone marrow aspiration procedure.
Sampling Method: Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Acceptance Criteria | Sample taken at initial visit with no follow up (Day 1)
  The acceptance criteria based on lower level of the 95% CI of the positive or negative percent agreement for all markers.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Tallman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Guido Marcucci, MD, Principal Investigator — James Cancer Hospital; Alan Burnett, MD, Principal Investigator — Cardiff University- School of Medicine; Hartmut Doehner, MD, Principal Investigator — University Hospital Ulm; Bob Lowenberg, MD, Principal Investigator — Erasmus Medical Center
Locations (5):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - James Cancer Hospital, Columbus, Ohio
- University Hospital Ulm, Ulm, Germany
- Erasmus Medical Center, Rotterdam, Netherlands
- Cardiff University, Cardiff, Heath Park, United Kingdom